CLINICAL TRIAL: NCT04301349
Title: Comparative Study Between Vaginal Dinoprostone and Vaginal Misoprostol Prior to IUD Insertion in Multiparous Women
Brief Title: Dinoprostone vs Misoprostol Before LNG-IUD Insertion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dinoprostone IUDs
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: IUD Insertion Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vaginal dinoprostone (Experimental): vaginal dinoprostone 6 mg (two tablets) 3 hours prior to IUD insertion
  Interventions: Drug: vaginal dinoprostone
- vaginal misoprostol (Active Comparator): vaginal misoprostol 400 mcg (two tablets) 3 hours prior to IUD insertion
  Interventions: Drug: vaginal misoprostol
- placebo (Placebo Comparator): two tablets of placebo similar in shape ,color, odor to the study drugs
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vaginal dinoprostone — two tablets of vaginal dinoprostone (6 mg) 3 hours prior to IUD insertion
  Arms: vaginal dinoprostone
Drug: vaginal misoprostol — two tablets of vaginal misoprostol (400 mcg) 3 hours prior to IUD insertion
  Arms: vaginal misoprostol
Drug: placebo — two tablets of placebo given 3 hours prior to IUD insertion
  Arms: placebo

SUMMARY:
the aim of this study is to compare the safety and efficacy of vaginal dinoprostone vs vaginal misoprostol administration prior to IUD insertion in multiparous women regarding reduction in iud insertion pain

ELIGIBILITY:
Inclusion Criteria:

* multiparous women requesting IUD insetion

Exclusion Criteria:

* active genital infection,uterine anomalies, and contraindication or allergy to dinoprostone or misoprostol

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
pain during IUD insertion: visual analog scale | 2 minutes
  pain during IUD insertion assessed by the visual analog scale from 0=no pain to 10 = the worst pain imaginable

SECONDARY OUTCOMES:
duration of IUD insertion | 5 minutes
  duration of IUD insertion measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, Principal Investigator — Cairo University